CLINICAL TRIAL: NCT06799832
Title: Urethral PeRfusion Index-Guided Hemodynamic ManagemenT in Patients Having Major Abdominal Surgery: the UPRIGHT Randomized Feasibility Trial
Acronym: UPRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-101408-BO-ff
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Urethral Perfusion Index; Tissue Perfusion; Microcirculation
Keywords: urethral perfusion index; tissue perfusion; microcirculation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine hemodynamic management (No Intervention): In patients assigned to routine hemodynamic management, hemodynamic management will be performed according to routine care. The urethral perfusion index measurements will not be visible.
- Urethral perfusion index guided hemodynamic monitoring (Experimental): In patients assigned to urethral perfusion index-guided hemodynamic monitoring, clinicians will be asked to maintaining the intraoperative urethral perfusion index above the postinduction baseline urethral perfusion index during surgery. Interventions to maintain intraoperative urethral perfusion index will be at the clinicians' discretion. All other medical procedures will be performed according to routine care. Clinical judgement will always prevail. Additionally, we will always strive to maintain macrocirculatory variables within predefined safety ranges: Mean arterial pressure: 60 mmHg - 120 mmHg Heart rate: 30 bpm - 120 bpm Cardiac index: at least 2.2 L/min/m2
  Interventions: Device: urethal perfusion index monitoring

INTERVENTIONS:
Device: urethal perfusion index monitoring — The urethral perfusion index will be monitored using the IKORUS System (Vygon, Écouen, France)
  Arms: Urethral perfusion index guided hemodynamic monitoring

SUMMARY:
We will perform this single-center pilot trial to determine if the intraoperative urethral perfusion index is higher in patients assigned to maintaining postinduction baseline urethral perfusion index than in patients assigned to routine care (with blinded urethral perfusion index monitoring). As pre-planned substudies, we will also assess the agreement between a) urethral perfusion index-derived pulse rate and heart rate measured with an electrocardiogram and b) between the urethral perfusion index and the peripheral perfusion index.

ELIGIBILITY:
Inclusion Criteria:

* at least 45 years old
* scheduled for elective major abdominal surgery (involving visceral organs with an expected duration of at least 120 minutes)
* indication for an arterial catheter
* indication for an urinary catheter

Exclusion Criteria:

* Pregnancy
* Planned surgery: nephrectomy, liver or kidney transplantation surgery
* Patients who previously had surgery on the urethra or bladder
* Patients without clinical indication for continuous blood pressure monitoring with an intraarterial catheter

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
average intraoperative urethral perfusion index | Start of surgery until end of surgery

SECONDARY OUTCOMES:
the absolute lowest intraoperative urethral perfusion index | Start of surgery until end of surgery
the lowest intraoperative 5-minute moving average urethral perfusion index | Start of surgery until end of surgery
the intraoperative area under the baseline urethral perfusion index | Start of surgery until end of surgery
the cumulative intraoperative duration with a urethral perfusion index below the baseline urethral perfusion index | Start of surgery until end of surgery
the percentage of surgical time the urethral perfusion index is above the postinduction baseline urethral perfusion index | Start of surgery until end of surgery
intraoperative area under a urethral perfusion index value 30% below baseline | Start of surgery until end of surgery
cumulative intraoperative duration with a urethral perfusion index below at least 30% lower than baseline | Start of surgery until end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, MD, Principal Investigator — University Medical Center Hamburg Eppendorf, Hamburg, Germany and OUTCOMES RESEARCH Consortium®, Houston, Texas, USA
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No